CLINICAL TRIAL: NCT07262346
Title: Clinical Pharmacokinetic Study of Hydronione Capsules in Healthy Chinese Subjects (Ⅰd)
Brief Title: The Phase Ⅰd Clinical Trial of Hydronidone Capsules
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDN-F351-202502
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Liver Fibrosis
Keywords: Hydronidone
MeSH Terms: conditions — Liver Cirrhosis | interventions — hydronidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- SAD:180mg drug group (Experimental): On the morning of D1, the patients took 180mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Hydronidone capsules
- SAD:120mg drug group (Experimental): On the morning of D1, the patients took 120mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Hydronidone capsules
- SAD:240mg drug group (Experimental): On the morning of D1, the patients took 240mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Hydronidone capsules
- SAD:300mg drug group (Experimental): On the morning of D1, the patients took 300mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Hydronidone capsules
- SAD:360mg drug group (Experimental): On the morning of D1, the patients took 360mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Hydronidone capsules
- SAD:420mg drug group (Experimental): On the morning of D1, the patients took 420mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Hydronidone capsules
- MAD: drug group1 (dosage to be determined) (Experimental): Single dose on an empty stomach on Days 1 and 8; on Days 2-7, take oral medication once every 8 hours.
  Interventions: Drug: Hydronidone capsules
- MAD: drug group 2 (dosage to be determined) (Experimental): Single dose on an empty stomach on Days 1 and 8; on Days 2-7, take oral medication once every 8 hours.
  Interventions: Drug: Hydronidone capsules
- MAD: drug group 3 (dosage to be determined) (Experimental): Single dose on an empty stomach on Days 1 and 8; on Days 2-7, take oral medication once every 8 hours.
  Interventions: Drug: Hydronidone capsules
- Study on the Interaction between Food and Drugs:drug group1 (dosage to be determined) (Experimental): Period 1 involved administration under fasting conditions, with a 7-day washout period starting on Day 2. Administration for Period 2 was conducted on Day 8.
  Interventions: Drug: Hydronidone capsules
- Study on the Interaction between Food and Drugs:drug group2 (dosage to be determined) (Experimental): In Period 1, a high-fat meal was consumed first, followed by drug administration within 30 minutes, with washout commencing on Day 2. After a total 7-day washout period, the second period of dosing was administered on Day 8.
  Interventions: Drug: Hydronidone capsules
- SAD:Placebo group (Placebo Comparator): On the morning of D1, the patients took 180mg of hydronidone capsules orally on an empty stomach once.
  Interventions: Drug: Placebo capsules
- MAD:Placebo group (Placebo Comparator): Single dose on an empty stomach on Days 1 and 8; on Days 2-7, take oral medication once every 8 hours.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Hydronidone capsules — SAD:Single-dose administration MAD:Multiple-dose group Study on the Interaction between Food and Drugs
  Arms: MAD: drug group 2 (dosage to be determined); MAD: drug group 3 (dosage to be determined); MAD: drug group1 (dosage to be determined); SAD:120mg drug group; SAD:180mg drug group; SAD:240mg drug group; SAD:300mg drug group; SAD:360mg drug group; SAD:420mg drug group; Study on the Interaction between Food and Drugs:drug group1 (dosage to be determined); Study on the Interaction between Food and Drugs:drug group2 (dosage to be determined)
Drug: Placebo capsules — SAD:Single-dose administration MAD:Multiple-dose group Study on the Interaction between Food and Drugs
  Arms: MAD:Placebo group; SAD:Placebo group

SUMMARY:
Based on the Phase I (Ia, Ib, Ic) clinical pharmacokinetic study of Hydronidone Capsules, a clinical pharmacokinetic trial of Hydronidone Capsules (specification: 30 mg/capsule) was conducted, including single-dose administration, multiple-dose administration, and a food-effect study. The aim was to investigate the safety, tolerability, and pharmacokinetic characteristics of higher doses of Hydronidone Capsules (specification: 30 mg/capsule) in healthy subjects, in preparation for future expansion of indications.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, both male and female;
2. Age: 18-45 years;
3. Weight: Male ≥50 kg, Female ≥45 kg, with a BMI between 19 and 26 (BMI = weight (kg)/height² (m²));
4. Pass a comprehensive health examination, meaning no abnormalities or no clinically significant findings in the following: vital signs, physical examination, blood and urine routine tests, blood pregnancy test, blood glucose, blood lipids, blood electrolytes, hepatitis B surface antigen, liver and kidney function, hepatitis C, HIV and syphilis antibody tests, 12-lead electrocardiogram, nicotine screening, urine drug screening, alcohol breath test, chest X-ray, etc.;
5. Have been fully informed about the nature, significance, potential benefits, possible inconveniences, and risks of the study prior to participation, and voluntarily agree to take part in this clinical trial. Subjects must be able to communicate well with the researchers, comply with all study requirements, and have the capacity to understand and sign the written informed consent form.

Exclusion Criteria:

1. (Inquiry) Participation in any other clinical trial within three months prior to this study;
2. (Inquiry) Presence of any disease that may affect the safety of the trial or the pharmacokinetics of the drug, including but not limited to: past or current diseases of the heart, liver, kidneys, endocrine system, digestive tract, immune system, respiratory system, nervous system, or psychiatric disorders [particularly cardiovascular diseases or individuals at risk of cardiovascular diseases, any gastrointestinal diseases affecting drug absorption (e.g., irritable bowel syndrome, inflammatory bowel disease), active pathological bleeding (e.g., peptic ulcer), urticaria, epilepsy, allergic rhinitis, eczematous dermatitis, asthma, active tuberculosis, etc.];
3. (Inquiry) Allergic constitution: such as a history of drug or food allergies, skin allergies, or lactose intolerance;
4. (Inquiry) Use of any drugs that inhibit or induce hepatic drug metabolism within 28 days before taking the investigational drug (common enzyme inducers: barbiturates such as phenobarbital, carbamazepine, aminoglutethimide, griseofulvin, meprobamate, phenytoin, glutethimide, rifampicin, dexamethasone; common enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamides);
5. Use of any medications (including herbal medicines) or health products within 14 days before the first dose;
6. (Inquiry) Individuals with special dietary requirements who cannot adhere to a standardized diet (e.g., intolerance to standard meals) or those with difficulty swallowing;
7. (Inquiry) Inability to tolerate venipuncture and/or a history of blood or needle phobia;
8. (Inquiry) Habitual excessive consumption of tea, coffee, or caffeine-containing beverages (more than 8 cups per day, 1 cup = 250 mL); or consumption of any caffeine-containing foods or beverages (e.g., coffee, strong tea, chocolate, etc.) within 48 hours before the first dose, or adherence to any special diet that may affect drug absorption, distribution, metabolism, or excretion;
9. (Inquiry) History of excessive alcohol consumption (defined as more than 28 standard units per week for men and more than 21 standard units per week for women (1 standard unit contains 14 g of alcohol, equivalent to 360 mL of beer, 45 mL of 40% spirits, or 150 mL of wine)); or regular alcohol consumption (more than 14 standard units per week) within 6 months prior to the trial; or consumption of any alcohol-containing products within 24 hours before the first dose;
10. (Inquiry) Blood donation or significant blood loss (exceeding 450 mL) within 3 months before the first dose, or plans to donate blood or blood components during the study or within 3 months after its completion;
11. (Inquiry) Occurrence of an acute illness during the pre-study screening phase or before administration of the study drug;
12. (Inquiry) Consumption of any foods or beverages known to induce or inhibit hepatic metabolic enzymes (e.g., grapefruit, mango, dragon fruit, grape juice, orange juice, etc., which are rich in flavonoids or citrus glycosides) within 24 hours before the first dose;
13. (Inquiry) Surgery within three months before screening or plans to undergo surgery during the study period;
14. (Inquiry) History of drug abuse or substance abuse;
15. (Inquiry) Smoking more than 5 cigarettes per day within 14 days before screening, or inability to discontinue the use of any tobacco products during the trial period;
16. (Inquiry) Smoking or use of any tobacco products between screening and hospital admission;
17. Positive nicotine test result;
18. Alcohol breath test result greater than 0.0 mg/100 mL;
19. Positive urine drug screen result;
20. Pregnant or breastfeeding women;
21. Individuals planning to conceive within 6 months after the trial or unwilling to use non-pharmacological contraceptive measures;
22. Any condition deemed by the investigator as potentially affecting the subject's ability to provide informed consent, comply with the trial protocol, or participate in the trial in a way that could impact the results or subject safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
SAD :Blood drug PK parameters(Cmax) | 24 hours after administration
SAD:Blood drug PK parameters（Tmax） | 24 hours after administration
SAD:Blood drug PK parameters（AUC0-t） | 24 hours after administration
SAD:Blood drug PK parameters( t1/2) | 24 hours after administration
SAD:Blood drug PK parameters(AUC0-∞) | 24 hours after administration
SAD:Blood drug PK parameters(λz) | 24 hours after administration
SAD:Blood drug PK parameters(Vd/F) | 24 hours after administration
SAD:Blood drug PK parameters(CL/F) | 24 hours after administration
SAD:Blood drug PK parameters(AUC_%Extrap) | 24 hours after administration
SAD:Blood drug PK parameters(MRT) | 24 hours after administration
MAD:Blood drug PK parameters(ss) | 24 hours after administration
MAD :Blood drug PK parameters(Cmax) | 24 hours after administration
MAD:Blood drug PK parameters（Tmax） | 24 hours after administration
MAD:Blood drug PK parameters（AUC0-t） | 24 hours after administration
MAD:Blood drug PK parameters( t1/2) | 24 hours after administration
MAD:Blood drug PK parameters(AUC0-∞) | 24 hours after administration
MAD:Blood drug PK parameters(λz) | 24 hours after administration
MAD:Blood drug PK parameters(Vd/F) | 24 hours after administration
MAD:Blood drug PK parameters(CL/F) | 24 hours after administration
MAD:Blood drug PK parameters(AUC_%Extrap) | 24 hours after administration
MAD:Blood drug PK parameters(MRT) | 24 hours after administration
The influence of food on the parameters of single-dose pharmacokinetics(Tlag) | 24 hours after administration
The influence of food on the parameters of single-dose pharmacokinetics(Cmax) | 24 hours after administration
The influence of food on the parameters of single-dose pharmacokinetics(Tmax) | 24 hours after administration
The influence of food on the parameters of single-dose pharmacokinetics(AUC0-t) | 24 hours after administration
The influence of food on the parameters of single-dose pharmacokinetics(AUC0-∞) | 24 hours after administration

SECONDARY OUTCOMES:
Hydronidone and its metabolites M3 and M4 blood drug concentrations (SAD) | 24 hours after administration
Hydronidone and its metabolites M3 and M4 blood drug concentrations (MAD) | 24 hours after administration
Safety indicator: Any adverse event | 48 hours after administration
  Adverse Event (AE) is defined as any untoward medical occurrence during drug clinical trials, drug therapy, or medical procedures, regardless of its causal relationship to the drug used.
Safety indicators:Chest X-ray examination | 48 hours after administration
Safety indicators:12-lead electrocardiogram examination. | 48 hours after administration
  The 12-lead electrocardiogram records the electrical activity of the heart through 12 different lead positions, and is the most commonly used and fundamental non-invasive examination method for diagnosing heart diseases.A 12-lead ECG examines P waves, PR intervals, QRS complexes, ST segments, T waves, QT intervals, and other ECG waves and intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China